CLINICAL TRIAL: NCT03297658
Title: Electro-acupuncture (EA) in Children Undergoing Procedures for Congenital Heart Defects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, David Rosen, MD, Principal Investigator, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1610318932
Record Dates: First submitted 2017-08-07; First posted 2017-09-29 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Congenital Heart Defect
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: All subjects will have electro-acupuncture pads applied at four points bilaterally: pericardial 4 (PC 4), pericardial 6 (PC 6), large intestine 4 (LI 4) and stomach 36 (ST 36). No needles will be used. (Appendix A; 1)
  Group 1: Receive electro-acupuncture (EA) (treatment) frequency will be at 2Hz and 100 Hz the amplitude will be microA.
  Group 2: Receive sham (control) will not have stimulation.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- electro-acupuncture (EA) intervention (Active Comparator): Micro electrodes will be placed at PC 4 and 6 , LI 4 and ST36. subjects will receive electro-acupuncture (EA) (treatment) mixed frequency( continuous plus dense disperse) will be at 2Hz and 100 Hz the amplitude will be 1000 microA.
  Interventions: Device: electro-acupuncture (EA)
- sham electro acupuncture (Sham Comparator): Micro electrodes will be placed at PC 4 and 6 , LI 4 and ST36. subjects Receive sham (control) will not have stimulation.
  Interventions: Device: sham

INTERVENTIONS:
Device: electro-acupuncture (EA) — stimulation of acupuncture points related to congenital heart surgery for comfort heart and renal health
  Arms: electro-acupuncture (EA) intervention
Device: sham — Micro electrodes will be placed but there will be no stimulation
  Arms: sham electro acupuncture

SUMMARY:
This is a single site, randomized, blinded, sham controlled, parallel group study to identify whether electro-acupuncture (EA) is a beneficial anesthesia adjunct in children undergoing procedures on their congenital heart defects (CHD).

DETAILED DESCRIPTION:
This investigation is a single site, randomized, blinded, sham controlled, parallel group study to identify whether EA is a beneficial anesthesia adjunct in children undergoing procedures on their congenital heart defects.

Study subjects age's birth to eighteen years, undergoing cardiac surgery for their congenital heart lesions will be considered for entrance into the study. The randomized subjects will receive either EA or sham during their surgery for CHD. Subjects are expected to remain in the hospital 48 hours post procedure. Standard of care blood samples will be obtained pre-operative and post-operative. The only study specific blood sample will be Troponin I levels which will be obtained before surgery begins after the IV lines have been placed, and 6 hours after bypass. Urine samples will be obtained before surgery after placement of the foley catheter and every 6 hours post bypass aortic cross clamp removal for 48 hours while the foley catheter is still in place.

ELIGIBILITY:
Inclusion Criteria:

* Patients 0-18 years of age undergoing procedures on their congenital heart defects where an aortic cross clamp will be placed.

Additionally, patients with coarctation of the aorta for repair will be considered as a separate group and eligible for enrollment.

* Willing to provide written Assent/Consent in English.

Exclusion Criteria:

* Patients with skin lesions over more than 50% of EA sites.
* Patients in renal failure.
* Patients on chronic opioid therapy.
* Unwilling to provide written Assent/Consent in English.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Change in Troponin level | baseline and 6 hours after weaning from cardiopulmonary bypass
  Troponin level Change from baseline. Troponin lab levels will be measured as a marker of myocardial injury. Children undergoing procedures for their congenital heart disease will have their troponin levels prior to the procedure and 6 hours after weaning from bypass. This study will look at differences between pre and post troponin values in the two groups.

SECONDARY OUTCOMES:
Evaluate the incidence and severity of pain in the post operative period | every 2 hours for 48 hours after arrival in Pediatric Intensive Care Unit (PICU)
  Subjects less than 2 month will have their pain assessed every 2 hours for 48 hours using the Neonatal Infant Pain Scale (NIPS).Pain in children 2 months to 7 years or those that are unable to communicate their pain will have their pain evaluated every 2 hours for 48 hours using the Face, Legs, Cry, Consolability Scale (FLACC). Scale range 0-10. Children older than 10 will have their pain evaluated every 2 hours for 48 hours using a Visual analogue scale (0-10).
Evaluate Acute Kidney Injury | baseline and 6,12,24, and 48 hours after weaning from Cardiopulmonary bypass
  Acute Kidney Injury (AKI) classification will be assessed using the AKIN classification system. This system uses Serum Creatinine and/or Urine output to come up with a staging of 1-3. Patients will be stage at 6, 12, 24, and 48 hours after bypass.

CONTACTS AND LOCATIONS:
Overall Officials: David A Rosen, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen DA, Unger K, Gustafson RA, Trieu C, Zeltzer LK, Lin YC. Electroacupuncture Addition to the Anesthesia Care of Pediatric Patients for Congenital Heart Surgery. J Cardiothorac Vasc Anesth. 2017 Aug;31(4):1497-1504. doi: 10.1053/j.jvca.2017.02.037. Epub 2017 Feb 8. No abstract available. PMID 28526209

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT03297658/Prot_SAP_000.pdf